CLINICAL TRIAL: NCT01933438
Title: Does Early Supination and External Rotation Repositioning in Children With Birth Related Brachial Plexus Injury Have Benefit? A Randomized Controlled Trial of the Sup-ER Protocol.
Brief Title: Sup-ER Protocol RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study ended early after encountering logistics challenges and difficulties with site recruitment.
Sponsor: University of British Columbia (Other)
Collaborators: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Cynthia Verchere, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H13-00751
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Birth Related Brachial Plexus Injury; Obstetrical Brachial Plexus Palsy
Keywords: birth related brachial plexus injury; brachial plexus; splint
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sup-ER protocol (Experimental): Early shoulder repositioning (Sup-ER Splint)
  Interventions: Other: Sup-ER Protocol
- Control (Active Comparator): Standard treatment
  Interventions: Other: Control

INTERVENTIONS:
Other: Sup-ER Protocol — Early shoulder repositioning (Sup-ER Splint)
  Arms: Sup-ER protocol
Other: Control — Standard treatment
  Arms: Control

SUMMARY:
This study evaluates the ability of a supination and external rotation protocol to improve the arm function and anatomy of children with birth related brachial plexus injuries.

DETAILED DESCRIPTION:
The brachial plexus is a group of 5 nerves from the spinal cord that provide the movement and sensation of an upper extremity. In some difficult deliveries, traction on the shoulder may lead to damage to the brachial plexus and will result in an arm that is paralyzed. This is called 'birth related brachial plexus injury' (BRBPI). This may occur in up to 1/1000 births and the nerves may be injured minimally to severely. About 2/3 of children with this injury will recover to quite functional levels simply by maintaining looseness of joints while their nerves slowly heal. Some children have nerve injuries severe enough that they require surgical reconstruction with nerve grafts and nerve transfers to achieve even adequate function. Even in children with otherwise "good" recovery, the motions of external rotation of the shoulder and supination of the forearm are weaker, later to recover, and often incomplete. More importantly, lack of full motion leads to long term changes in the structure, growth, and posture of the shoulder requiring further musculoskeletal surgery, or a child with permanent deformity or disability.

Any gains in active and passive range of motion during the first year of life may improve these long-term shoulder outcomes. The investigators have instituted a program of early passive repositioning mostly using a custom Sup-ER (Supination and External Rotation) splint during early growth and development to improve arm position and range of motion where ER and Sup are weak. In compliant patients in a pilot study, the speed and strength of recovery of ER and Supination are improved compared to historical controls. It is a novel splint and protocol designed by the investigators. This study is a randomized controlled trial to evaluate the use of the Sup-ER protocol in multiple centres over a two year period by assessing the arm function at common time points in recovery. The subjects are randomized to the Sup-ER protocol or the currently accepted standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brachial plexus injury at birth.
* Significant deficit in external rotation and/or supination of the affected limb based on clinical assessment using the Toronto Active Movement Scale at 6 weeks of age (External Rotation ≤ 2 and/or Supination ≤ 2)
* Tightness in Passive Range of Motion of external rotation: any angle of less than 180°.
* Age 6-8 weeks

Exclusion Criteria:

* Neuromuscular disorder
* Unwillingness or inability to comply with the requirements of the study protocol.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Toronto Active Movement Scale | 1 year of age

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Verchere, MD FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada